CLINICAL TRIAL: NCT07381530
Title: A Prospective Randomized, Single-blind, Multicenter Phase II Study Comparing Two Methods of Cardioplegia in Cardiac Surgery Due to Congenital Heart Malformation in Children: Custodiol-N Versus Custodiol
Brief Title: Study of Cardioplegia in Cardiac Surgery Due to Congenital Heart Malformation in Children
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Dr. F. Köhler Chemie GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL-N-CP-Paed-II/09/19
Record Dates: First submitted 2024-10-28; First posted 2026-02-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Congenital Heart Malformations
MeSH Terms: interventions — Custodiol-N solution

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient and their legal representatives will be blinded to treatment. All other parties are unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custodiol-N (Experimental): organ will be perfused with Custodiol-N solution
  Interventions: Drug: heart will be treated with Custodiol-N
- Custodiol (Active Comparator): organ will be perfused with Custodiol solution
  Interventions: Drug: heart will be treated with Custodiol

INTERVENTIONS:
Drug: heart will be treated with Custodiol-N — cardioplegia solution will be administered with perfusion
  Arms: Custodiol-N
Drug: heart will be treated with Custodiol — cardioplegia solution will be administered with perfusion
  Arms: Custodiol

SUMMARY:
The objective of this investigation is to compare the safety and cardioprotective effects of Custodiol and Custodiol-N in children undergoing cardiac surgery with cardiopulmonary bypass (CPB) due to congenital heart malformation. All endpoint timings refer to the opening of the aortic cross clamp (t=0)

DETAILED DESCRIPTION:
Efficacy of Custodiol-N and its safety is being thoroughly studied in adults undergoing solid organ transplantation. In addition, safety data are available from its use as cardioplegic solution in approximately 400 adults. Paediatric cardiac surgery nearly exclusively addresses congenital heart disease (CHD). CHD comprises a wide variety of congenital malformations of structures of the heart or the great vessels. The causes may be genetic, environmental or both. The objective of this investigation is to compare the safety and cardioprotective effects of Custodiol and Custodiol-N in children undergoing cardiac surgery with cardiopulmonary bypass (CPB) due to congenital heart malformation.

ELIGIBILITY:
Inclusion Criteria:

* Age from birth to less than 18 years of age
* congenital heart surgery with cardiopulmonary bypass and cardioplegia
* written informed consent of the patients and/ or their legal guardians (must be available before enrolment in the study)
* Ability of the legal guardians to understand character and individual consequences of the clinical trial

Exclusion Criteria:

* Patients who have participated within 30 days or are still participating in any other interventional study
* History of severe organic (e.g. liver or kidney) disease other than concerning the heart
* History of psychiatric disease
* Pregnancy and lactation

Ages: 24 Hours to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
safety assessment | AEs up to 30 days postoperatively
  Continuous adverse events (AEs) reporting
safety assessment | CK-MB (Creatinkinase-MB) levels at baseline until postoperative day 2 and postoperative day 7 or discharge
  Myocardial protection in surviving patients assessed by quantification of perioperative CK-MB levels (U/l)

SECONDARY OUTCOMES:
Description of hemodynamics | day 7 postoperatively
  Vital signs (blood pressure (mmHg))
Description of hemodynamics | day 7 postoperatively
  Vital signs (heart rate (bpm))
Description of hemodynamics | day 7 postoperatively
  Vital signs (body temperature (°C))
Description of hemodynamics | day 7 postoperatively
  Vasopressor/ Catecholamine/ Vasodilator (incl. Milrinone)/ Levosimendan intake (yes/no by timepoint and amount (μg/kg/min))
Description of hemodynamics | day 7 postoperatively
  Nitric oxide ventilation (yes/no by timepoint)
Description of hemodynamics | day 7 postoperatively
  Extracorporeal membrane oxygenation (ECMO) support (yes/no by timepoint)
Description of hemodynamics | 30 days postoperatively
  Need for placement of a permanent Medical Circulatory Support (MCS) (left ventricular assist device (LVAD), right ventricular assist device (RVAD), biventricular assist support (BiVAD)), (yes/no by timepoint)
Description of hemodynamics | 30 days postoperatively
  Need for heart transplant (yes/no by timepoint)
Description of echo | Baseline, after skin closure and day 7 postoperatively
  Systemic-ventricular function (good, moderately impaired, severely impaired)
Description of cardiac injury | at baseline until postoperative day 2 and postoperative day 7 or discharge
  Creatine kinase (CK (U/l))
Description of cardiac injury | at baseline until postoperative day 2 and postoperative day 7 or discharge
  Troponin T (ng/ml)
Description of hospitals stay/ death | 30 days postoperatively
  Death (date)
Description of hospitals stay/ death | 30 days postoperatively
  readmission (to hospital or intensive care), (yes/no and number)
Description of hospitals stay/ death | 30 days postoperatively
  Length of ICU stay (start and end date)
Description of hospitals stay/ death | 30 days postoperatively
  Length of hospital stay (start and end date)
Description of surgery | during surgery
  Aortic cross clamping time (min)
Description of surgery | during surgery
  Incision-to-closure-time (min)
Description of surgery | during surgery
  Reperfusion time (min)
Description of surgery | during surgery
  Number of intraoperative administrations of cardioplegia
Description of surgery | during surgery
  Total administration duration (min)
Description of surgery | during surgery
  Total administration amount (ml)
Description of 12-Lead-ECG | baseline and day 1 postoperatively (Intensive Care Unit)
  Shift in 12-Lead-ECG (ECG QT Interval)
Description of cardiac arrhythmias | until day 7 postoperatively
  Current heart rhythm (Sinus rhythm, atrioventricular block (AV-Block °I), AV-Block °II, AV-Block °III, Ectopic atrial rhythm with intact AV conduction, other tachycardiac arrhythmia)
Description of cardiac arrhythmias | until day 7 postoperatively
  Tachyarrhythmic event since last visit (JET/atrial fibrillation/atrial flutter/ ventricular arrhythmia)
Description of cardiac arrhythmias | until day 7 postoperatively
  Need for antiarrhythmic therapy other than beta blockers after end of aortic cross-clamping since last visit (e.g. Adenosine, Amiodarone, Flecainid), (yes/no)
Description of cardiac arrhythmias | 30 days postoperatively
  Current cardiac pacing (none/atrial/ventricular/sequential)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Grieshaber, PD Dr., Principal Investigator — Sektion Kinderherzchirurgie, Klinik für Herz- und Thoraxchirurgie, Universitätsklinikum Münster, Germany; Christine-Elena Kamla, Dr., Principal Investigator — Deutsches Herzzentrum München, TUM Universitätsklinikum, Germany; Mohamed Salem, Dr., Principal Investigator — Kinderherzzentrum, Universitätsklinikum Gießen und Marburg GmbH, Germany
Locations (3):
- Germany (3):
  - Universitätsklinikum Gießen und Marburg GmbH, Abteilung für Kinderherzchirurgie und angeborene Herzfehler, Giessen
  - Deutsches Herzzentrum München, TUM Universitätsklinikum, Klinik für Chirurgie angeborener Herzfehler und Kinderherzchirurgie, München
  - Universitätsklinikum Münster, Klinik für Herz- und Thoraxchirurgie,Sektion Kinderherzchirurgie, Münster

IPD SHARING:
Plan to Share IPD: No